CLINICAL TRIAL: NCT07184177
Title: Validation of the Accuracy of Heart Rate Monitors at Resting and Exercise at Maximal Fat Oxidation Rate in Overweight and Obese Young Adults
Brief Title: Validation of Heart Rate Monitors in Overweight and Obese Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Marco Antonio Hernández Lepe, Full Time Professor, Universidad Autonoma de Baja California
Other Study IDs: Validation Heart Rate Monitors
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation group: Participants to validate 10 heart rate monitors against electrocardiogram at resting and exercise at a maximal fat oxidation rate

SUMMARY:
Overweight and obesity are defined as an excessive accumulation of body fat that affects health. According to data from the World Health Organization (WHO), in 2022, there were 2.5 billion adults aged 18 years and older who were overweight, of whom 890 million were obese. In other words, 43% of adults aged 18 years and older were overweight, and 16% of them were obese.

Overweight and obesity are key risk factors for various chronic diseases such as diabetes, hypertension, cardiovascular disease, and even some types of cancer. There is evidence that mortality from cardiovascular disease, and the incidence of cancer and diabetes, varies according to the amount of physical activity. In the context of high levels of sedentary time, higher levels of moderate to vigorous physical activity are recommended. There are various ways to treat overweight and obesity, the main ones usually being lifestyle changes, such as following a healthy diet and regular physical activity, as well as following pharmacological treatments. In this project, the focus will be on the fat metabolism generated during moderate physical activity.

There are physical activity interventions aimed at increasing fat metabolism that may potentially reduce the symptoms of metabolic diseases such as obesity and type 2 diabetes. For this purpose, it is important to understand the factors that increase or decrease fat oxidation. Factors such as exercise intensity and duration are important to understand when determining maximum fat oxidation (FatMax).

The aim is to develop comprehensive research that will generate knowledge and evidence on health issues with social impact through the evaluation of commercial technologies and innovative actions that promote the prevention, treatment, and resolution of national health problems such as obesity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 25 kg/m2
* Energy expenditure < 600 METs a week
* Acceptance of informed consent

Exclusion Criteria:

* ≥100 mL of alcohol consumption per week
* Have limitations to perform regular physical activity
* Have a chronic non-communicable disease
* Answer "yes" to any of the questions on the Physical Activity Readiness-Questionnaire for Everyone (PAR-Q+), which represents a health risk.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sedentary young adults aged between 18 and 35 years, all of whom will have a body mass index (BMI) ≥ 25 kg/m2. Participants will be recruited through snowball sampling.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Heart rate at maximal fat oxidation | 30 minutes
  Gas exchange and heart rate will be recorded throughout the exercise tests, while the rate of perceived exertion will be registered at the end of each stage using the modified Borg scale with a 0-10 rating. The average VO2 and VCO2 values of the last 2 min of each stage before RER ≥ 1.0 will be used to calculate fat and carbohydrate oxidation using the stoichiometric equations of Jeukendrup and Wallis. The maximum rate of fat oxidation and its corresponding intensity during exercise will be determined by mathematical modeling of fat oxidation kinetics, plotted against oxygen consumption (% VO2max). The symmetry, amplitude, and translation parameters of the curve will be calculated as well to represent the oxidative capacity of each subject.
Resting heart rate | 30 minutes
  Resting heart rate of participants using 10 different heart rate monitors

IPD SHARING:
Plan to Share IPD: Yes
Publication of original article in an indexed journal with impact factor (JCR) over 2.0.

REFERENCES:
- [Background] Chavez-Guevara IA, Amaro-Gahete FJ, Ramos-Jimenez A, Brun JF. Toward Exercise Guidelines for Optimizing Fat Oxidation During Exercise in Obesity: A Systematic Review and Meta-Regression. Sports Med. 2023 Dec;53(12):2399-2416. doi: 10.1007/s40279-023-01897-y. Epub 2023 Aug 16. PMID 37584843
- [Background] Hernandez-Lepe MA, Hernandez-Ontiveros DA, Chavez-Guevara IA, Ramos-Jimenez A, Hernandez-Torres RP, Lopez-Fregoso RJ, Ramos-Lopez O, Amaro-Gahete FJ, Muniz-Salazar R, Olivas-Aguirre FJ. Impact of Exercise Training at Maximal Fat Oxidation Intensity on Metabolic and Epigenetic Parameters in Patients with Overweight and Obesity: Study Protocol of a Randomized Controlled Trial. J Funct Morphol Kinesiol. 2024 Oct 31;9(4):214. doi: 10.3390/jfmk9040214. PMID 39584867
- [Background] Chavez-Guevara IA, Urquidez-Romero R, Perez-Leon JA, Gonzalez-Rodriguez E, Moreno-Brito V, Ramos-Jimenez A. Chronic Effect of Fatmax Training on Body Weight, Fat Mass, and Cardiorespiratory Fitness in Obese Subjects: A Meta-Analysis of Randomized Clinical Trials. Int J Environ Res Public Health. 2020 Oct 28;17(21):7888. doi: 10.3390/ijerph17217888. PMID 33126461